CLINICAL TRIAL: NCT05594589
Title: A Multicenter, Double-Blind, Randomized, Placebo-Controlled, Parallel-Group Study to Assess the Pharmacodynamics of Lemborexant in Korean Subjects With Insomnia Disorder
Brief Title: A Study to Assess the Pharmacodynamics of Lemborexant in Korean Participants With Insomnia Disorder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eisai Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Eisai Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: E2006-J082-204
Record Dates: First submitted 2022-10-21; First posted 2022-10-26 (Actual); Results first posted 2025-07-03 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-05

CONDITIONS: Sleep Initiation and Maintenance Disorders
Keywords: Lemborexant; E2006; Dayvigo
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — lemborexant

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Lemborexant 5 mg (LEM5) (Experimental): Participants will receive one LEM5 tablet, orally, once daily for 30 nights (Day 1 up to Day 30) on each night approximately 5 minutes before participants intend to try to sleep.
  Interventions: Drug: Lemborexant
- Lemborexant 10 mg (LEM10) (Experimental): Participants will receive one lemborexant 10 mg (LEM10) tablet, orally, once daily for 30 nights (Day 1 up to Day 30) on each night approximately 5 minutes before participants intend to try to sleep.
  Interventions: Drug: Lemborexant
- Placebo (PBO) (Placebo Comparator): Participants will receive one lemborexant-matched PBO tablet, orally, once daily for 30 nights (Day 1 to Day 30) on each night approximately 5 minutes before participants intend to try to sleep.
  Interventions: Other: PBO

INTERVENTIONS:
Drug: Lemborexant — Lemborexant oral tablet.
  Other Names: E2006; Dayvigo
  Arms: Lemborexant 10 mg (LEM10); Lemborexant 5 mg (LEM5)
Other: PBO — Lemborexant-matched PBO tablet.
  Arms: Placebo (PBO)

SUMMARY:
The primary purpose of the study is to evaluate the treatment difference between lemborexant 5 milligram (mg) (LEM5) and placebo (PBO) on latency to persistent sleep (LPS) using polysomnography (PSG) on Day 30.

ELIGIBILITY:
Inclusion Criteria:

1. Korean male or female, age 19 to 80 years, at the time of informed consent
2. Meets the Diagnostic and Statistical Manual of Mental Disorders, 5th Edition (DSM-5) criteria for Insomnia Disorder, as follows:

   * Complains of dissatisfaction with nighttime sleep, in the form of difficulty getting to sleep with or without difficulty staying asleep and/or awakening earlier in the morning than desired despite adequate opportunity for sleep
   * Frequency of complaint greater than or equal to (>=) 3 times per week
   * Duration of complaint >= 3 months
   * Associated with complaint of daytime impairment
3. Subjective Sleep Onset Latency (sSOL) typically >= 30 minutes on at least 3 nights per week in the previous 4 weeks at Screening
4. Insomnia Severity Index (ISI) score >=13 at Screening
5. Regular time in bed between 6.5 and 9.0 hours at Screening
6. At 2nd Screening Visit (Visit 2): Confirmation (via Sleep Diary) of a regular bedtime, defined as the time the participant attempts to sleep, between 21:00 and 24:00 on at least 5 of the final 7 nights and regular waketime, defined as the time the participant gets out of bed for the day, between 05:00 and 09:00 on at least 5 of the final 7 nights.
7. Confirmation of current insomnia symptoms, as determined from responses on the sleep diary on the 7 most recent mornings before the PSG during Screening Period (Visit 2), such that sSOL >=30 minutes on at least 3 of the 7 nights
8. Confirmation of sufficient duration of time spent in bed, as determined from responses on the sleep diary on the 7 most recent mornings before the 2nd Screening Visit (Visit 2), such that there are no more than 2 nights with time spent in bed duration less than (<) 7 hours or greater than (>) 10 hours
9. During Run-in period, objective (PSG) evidence of insomnia as follows:

   * SE less than or equal to (<=) 85 percent (%); and
   * LPS >= 30 minutes
10. Provide written informed consent
11. Willing and able to comply with all aspects of the protocol, including staying in bed for at least 7 hours each night

Exclusion Criteria:

1. Females who are breastfeeding or pregnant at Screening or Baseline (as documented by a positive beta-human chorionic gonadotropin (beta-hCG). A separate baseline assessment is required if a negative screening pregnancy test was obtained more than 72 hours before the 1st dose of study drug
2. Females of childbearing potential who:

   * Within 28 days before study entry, did not use a highly effective method of contraception, which includes any of the following:

     * total abstinence (if it is their preferred and usual lifestyle)
     * an intrauterine device or intrauterine hormone-releasing system (IUS)
     * a contraceptive implant
     * an oral contraceptive (Participant must have been on a stable dose of the same oral contraceptive product for at least 28 days before dosing and must agree to stay on the same dose of the oral contraceptive throughout the study and for 28 days after study drug discontinuation.)
     * have a vasectomized partner with confirmed azoospermia
   * Do not agree to use a highly effective method of contraception (as described above) throughout the entire study period and for 28 days after study drug discontinuation. It is permissible that if a highly effective method of contraception is not appropriate or acceptable to the participant, then the participant must agree to use a medically acceptable method of contraception, that is, double-barrier methods of contraception such as latex or synthetic condom plus diaphragm or cervical/vault cap with spermicide NOTE: All females will be considered to be of childbearing potential unless they are postmenopausal (amenorrheic for at least 12 consecutive months, in the appropriate age group, and without other known or suspected cause) or have been sterilized surgically (that is, bilateral tubal ligation, total hysterectomy, or bilateral oophorectomy, all with surgery at least 1 month before dosing)
3. Any history of a medical or psychiatric condition that in the opinion of the investigator(s) could affect the participants safety or interfere with the study assessments
4. A prolonged QT interval corrected for heart rate by Fridericia's formula (QTcF) interval (QTcF >450 millisecond [ms]) as demonstrated by a repeated ECG. A history of risk factors for torsade de pointes (example, heart failure, hypokalemia, family history of long QT Syndrome) or the use of concomitant medications that prolonged the QTcF interval
5. Any suicidal ideation with intent with or without a plan at Screening or within 6 months of Screening
6. Any lifetime suicidal behavior
7. Evidence of clinically significant disease (example, cardiac; respiratory including chronic obstructive pulmonary disease, acute and/or severe respiratory depression; gastrointestinal; moderate and severe hepatic impairment; renal including severe renal impairment; neurological including myasthenia gravis; psychiatric disease; or malignancy within the past 5 years other than adequately treated basal cell carcinoma) or chronic pain that in the opinion of the investigator(s) could affect the participants safety or interfere with the study assessments. Participants for whom a sedating drug would be contraindicated for safety reasons because of the participants occupation or activities
8. Hypersensitivity to lemborexant or to their excipients
9. Scheduled for surgery during the study that requires general anesthesia or administration of prohibited medications
10. Known to be human immunodeficiency virus (HIV) positive
11. Active viral hepatitis (B or C) as demonstrated by positive serology
12. History of drug or alcohol dependency or abuse within approximately the last 2 years
13. A current diagnosis of sleep-related breathing disorder including obstructive sleep apnea (with or without continuous positive airway pressure [CPAP] treatment), periodic limb movement disorder, restless legs syndrome, circadian rhythm sleep disorder, or narcolepsy, or an exclusionary score on screening instruments to rule out individuals with symptoms of certain sleep disorders other than insomnia as follows:

    * STOPBang score >=5
    * International Restless Legs Scale (IRLS) >=16
14. Apnea-Hypopnea Index >15 or Periodic Limb Movement with Arousal Index >15 as measured on the PSG at the 2nd Screening Visit
15. Reports symptoms potentially related to narcolepsy, that in the clinical opinion of the investigator indicates the need for referral for a diagnostic evaluation for the presence of narcolepsy
16. Reports a history of sleep-related violent behavior, or sleep driving, or any other complex sleep-related behavior (example, making phone calls or preparing and eating food while sleeping)
17. For participants who underwent diagnostic PSG within 1 year before informed consent:

    * Age 19 to 64 years: Apnea hypopnea Index >=10, or Periodic Limb Movements with Arousal Index >=10,
    * Age >=65 years: Apnea Hypopnea Index >15, or Periodic Limb Movements with Arousal Index >15
18. Beck Depression Inventory-II (BDI-II) score >19 at Screening
19. Beck Anxiety Inventory (BAI) score >15 at Screening
20. Habitually naps during the day more than 3 times per week
21. Excessive caffeine use that in the opinion of the investigator contributes to the participants insomnia, or habitually consumes caffeine containing beverages after 18:00 and is unwilling to forego caffeine after 18:00 for the duration of his/her participation in the study. Participants are excluded if, in the previous 3 months, they had symptoms that would meet DSM-5 criteria for caffeine intoxication, which includes consumption of a high dose of caffeine (significantly in excess of 250 mg) and >=5 of the following symptoms: restlessness, nervousness, excitement, insomnia, flushed face, diuresis, gastrointestinal disturbance, muscle twitching, rambling flow of thought and speech, tachycardia or cardiac arrhythmia, periods of high energy, or psychomotor agitation. To be exclusionary, those symptoms must cause distress or impairment in social, occupational and other forms of functioning, and not be associated with other substance, mental disorder or medical condition
22. Reports habitually consuming more than 14 drinks containing alcohol per week (females) or more than 21 drinks containing alcohol per week (males), or unwilling to limit alcohol intake to no more than 2 drinks per day or forego having alcohol within the 3 hours before bedtime for the duration of his/her participation in the study
23. Comorbid nocturia that is causing or exacerbating the insomnia
24. Used any prohibited prescription or over-the-counter concomitant medications within 1 week or 5 half-lives, whichever is longer, before the 1st dose of study medication (Run-in Period)
25. Used any modality of treatment for insomnia, including cognitive behavioral therapy or marijuana within 1 week or 5 half-lives, whichever is longer, before the 1st dose of study medication (Run-in Period)
26. Failed treatment with dual orexin receptor antagonist drugs (efficacy and/or safety) following treatment with an appropriate dose and of adequate duration in the opinion of the investigator
27. Transmeridian travel across more than 3 time zones in the 2 weeks before Screening, or between Screening and Baseline, or plans to travel across different time zones during the study
28. Performed shift work in the 2 weeks before Screening, or between Screening and Baseline, or plans to do during the study
29. A positive drug test at Screening, Run-in, or Baseline, or unwilling to refrain from use of recreational drugs during the study
30. Currently enrolled in another clinical trial or used any investigational drug or device within 30 days or 5* the half-life, whichever is longer, preceding informed consent
31. Previously participated in any clinical trial of lemborexant

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2022-11-30 (Actual); Primary Completion 2024-04-26 (Actual); Study Completion 2024-05-24 (Actual)

CONTACTS AND LOCATIONS:
Locations (9):
- South Korea (9):
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - The Catholic University of Korea, St. Vincent Hospital, Suwon, Gyeonggi-do
  - Keimyung University Dongsan Hospital, Daegu
  - Gacheon University Gil Medical Centre, Incheon
  - Seoul National University Hospital, Seoul
  - Konkuk University Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - Korea University Guro Hospital, Seoul
  - Kyung Hee University Hospital at Gangdong, Seoul

IPD SHARING:
Plan to Share IPD: Yes
Eisai's data sharing commitment and further information on how to request data can be found on our website http://eisaiclinicaltrials.com/.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 9 investigative sites in South Korea from 30 November 2022 to 24 May 2024.
Pre-assignment Details: A total of 183 participants were screened, of which 118 were screen failure, and 65 participants received placebo in Run-in Period. Participants who completed Run-in period were randomized in Treatment Period to receive placebo, lemborexant 5 milligrams (mg) or lemborexant 10 mg.
Groups:
- Placebo: Participants received one lemborexant-matched placebo tablet, orally, once daily, approximately 5 minutes before intend to sleep for 30 nights from Day 1 up to Day 30 in Treatment Period.
- Lemborexant 5 mg: Participants received one lemborexant 5 mg tablet, orally, once daily, approximately 5 minutes before intend to sleep for 30 nights from Day 1 up to Day 30 in Treatment Period.
- Lemborexant 10 mg: Participants received one lemborexant 10 mg tablet, orally, once daily, approximately 5 minutes before intend to sleep for 30 nights from Day 1 up to Day 30 in Treatment Period.
Period: Overall Study
Arm/Group | Placebo | Lemborexant 5 mg | Lemborexant 10 mg
Started | 13 | 26 | 26
Treated During Treatment Period | 13 | 26 | 26
Placebo Run-in Period (Participants received one lemborexant-matched PBO tablet, orally, once daily, approximately 5 minutes before intend to sleep for 14 nights from Day -14 up to Day 1 (Baseline) during Run-in Period.) | 65 | 0 | 0
Completed | 13 | 25 | 26
Not Completed | 0 | 1 | 0
Not completed — Other | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: The safety analysis set included participants who received at least 1 dose of randomized study drug and had at least 1 post-dose safety assessment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Lemborexant 5 mg | Lemborexant 10 mg | Total
Number analyzed (Participants) | 13 | 26 | 26 | 65
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 12 | 20 | 25 | 57
  >=65 years | 1 | 6 | 1 | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.6 (13.33) | 49.1 (15.85) | 43.2 (13.84) | 46.2 (15.03)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 13 | 17 | 40
  Male | 3 | 13 | 9 | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 13 | 26 | 26 | 65
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 13 | 26 | 26 | 65
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Treatment Period: Change From Baseline in Latency to Persistent Sleep (LPS) on Day 30 of Lemborexant 5 mg Compared to Placebo
Description: LPS is the duration of time measured from lights off to the first epoch of 20 consecutive epochs of non-wakefulness as measured by polysomnography (PSG).
Time Frame: Baseline, at Day 30
Population: The full analysis set (FAS) included the group of randomized participants who received at least 1 dose of randomized study drug and had LPS data from the PSG on Day 30.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Placebo | Lemborexant 5 mg
Number analyzed (Participants) | 13 | 25
minutes | -46.12 (59.006) | -50.90 (55.263)
Statistical Analysis 1: Comparison: Placebo vs Lemborexant 5 mg; Test type: Superiority; p = 0.0133, ANCOVA; P-value was based on analysis of covariance (ANCOVA) model with log transformation of baseline LPS and treatment arms as fixed effects; Least Squares Geometric Mean(LSGM) Ratio = 0.377, 95% CI 2-sided [0.175 to 0.810] — LSGM ratio was calculated as Lemborexant 5 mg/Placebo

2. Secondary Outcome: Treatment Period: Change From Baseline in LPS on Day 30 of Lemborexant 10 mg Compared to Placebo
Description: LPS is the duration of time measured from lights off to the first epoch of 20 consecutive epochs of non-wakefulness as measured by PSG.
Time Frame: Baseline, at Day 30
Population: The FAS included the group of randomized participants who received at least 1 dose of randomized study drug and had LPS data from the PSG on Day 30.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Placebo | Lemborexant 10 mg
Number analyzed (Participants) | 13 | 26
minutes | -46.12 (59.006) | -44.15 (68.632)
Statistical Analysis 1: Comparison: Placebo vs Lemborexant 10 mg; Test type: Superiority; p = 0.0619, ANCOVA; P-value was based on ANCOVA model with log transformation of baseline LPS and treatment arms as fixed effects; LSGM Ratio = 0.480, 95% CI 2-sided [0.222 to 1.038] — LSGM ratio was calculated as Lemborexant 10 mg/Placebo

3. Secondary Outcome: Treatment Period: Change From Baseline in Objective Sleep Efficiency (SE) on Day 30 of Lemborexant 5 mg Compared to Placebo
Description: SE is defined as total sleep time (TST) divided by time spent in bed multiplied by 100 as measured by PSG. TST is duration of sleep from sleep onset until terminal awakening.
Time Frame: Baseline, at Day 30
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentage of time in bed asleep
Arm/Group | Placebo | Lemborexant 5 mg
Number analyzed (Participants) | 13 | 25
percentage of time in bed asleep | 8.32 (14.730) | 15.06 (12.292)
Statistical Analysis 1: Comparison: Placebo vs Lemborexant 5 mg; Test type: Superiority; p = 0.0689, ANCOVA; P-value was based on ANCOVA model with log transformation of baseline LPS and treatment arms as fixed effects; Least Square Mean (LSM) Difference = 7.38, 95% CI 2-sided [-0.59 to 15.35] — LSM difference was calculated as Lemborexant 5 mg - Placebo

4. Secondary Outcome: Treatment Period: Change From Baseline in Objective SE on Day 30 of Lemborexant 10 mg Compared to Placebo
Description: SE is defined as TST divided by time spent in bed multiplied by 100 as measured by PSG. TST is duration of sleep from sleep onset until terminal awakening.
Time Frame: Baseline, at Day 30
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentage of time in bed asleep
Arm/Group | Placebo | Lemborexant 10 mg
Number analyzed (Participants) | 13 | 26
percentage of time in bed asleep | 8.32 (14.730) | 15.44 (13.160)
Statistical Analysis 1: Comparison: Placebo vs Lemborexant 10 mg; Test type: Superiority; p = 0.0439, ANCOVA; P-value was based on ANCOVA model with log transformation of baseline LPS and treatment arms as fixed effects; LSM Difference = 8.16, 95% CI 2-sided [0.23 to 16.09] — LSM difference was calculated as Lemborexant 10 mg - Placebo

5. Secondary Outcome: Treatment Period: Number of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: A TEAE was defined as an adverse event (AE) that emerges during treatment (on or after the first dose of study drug up to 28 days after the participant's last dose), having been absent at pretreatment (Baseline) or reemerges during treatment, having been present at pretreatment but stopped before treatment, or worsens in severity during treatment relative to the pretreatment state, when the AE was continuous.
Time Frame: From start of study drug administration at Day 1 up to Day 58
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Lemborexant 5 mg | Lemborexant 10 mg
Number analyzed (Participants) | 13 | 26 | 26
Participants | 1 | 5 | 2

6. Secondary Outcome: Treatment Period: Number of Participants With Clinically Significant Abnormal Laboratory Parameters
Description: The laboratory parameters included hematology, chemistry, and urinalysis. Any abnormality in the laboratory results which are deemed clinically significant by the investigator were reported.
Time Frame: From start of study drug administration at Day 1 up to Day 58
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Lemborexant 5 mg | Lemborexant 10 mg
Number analyzed (Participants) | 13 | 26 | 26
Participants | 0 | 0 | 0

7. Secondary Outcome: Treatment Period: Number of Participants With Clinically Significant Abnormal Vital Signs Values
Description: Vital sign measurement included systolic and diastolic blood pressure, pulse rate, respiratory rate and body temperature. Any abnormality in vital signs which are deemed clinically significant by the investigator were reported.
Time Frame: From start of study drug administration at Day 1 up to Day 58
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Lemborexant 5 mg | Lemborexant 10 mg
Number analyzed (Participants) | 13 | 26 | 26
Participants | 0 | 0 | 0

8. Secondary Outcome: Treatment Period: Number of Participants With Clinically Significant Abnormal Electrocardiograms (ECGs) Findings
Description: Any abnormality in ECG assessments which were deemed clinically significant by the investigator were reported.
Time Frame: From start of study drug administration at Day 1 up to Day 58
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Lemborexant 5 mg | Lemborexant 10 mg
Number analyzed (Participants) | 13 | 26 | 26
Participants | 0 | 0 | 0

9. Secondary Outcome: Treatment Period: Plasma Concentrations of Lemborexant and Its Metabolites (M4, M9, and M10)
Description: Plasma concentrations of lemborexant and its metabolites M4, M9, and M10 were reported.
Time Frame: Within 2 hours pre-dose on Day 30; At 1 and 1.5 hours after morning waketime on Day 31
Population: The pharmacokinetic (PK) analysis set included the group of participants who had at least 1 quantifiable plasma concentration of lemborexant or its metabolites, with adequately documented dosing history.
Measure: Mean (Standard Deviation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Lemborexant 5 mg | Lemborexant 10 mg
Number analyzed (Participants) | 24 | 26
nanogram per milliliter (ng/mL)
  Lemborexant, Day 30: Pre-dose | 4.00 (6.20) | 9.13 (10.3)
  M4, Day 30: Pre-dose | 2.10 (2.68) | 5.60 (5.87)
  M9, Day 30: Pre-dose | 0.501 (0.622) | 1.33 (1.48)
  M10, Day 30: Pre-dose | 1.86 (2.22) | 5.43 (5.51)
  Lemborexant, Day 31: At 1 hour after morning waketime | 7.72 (4.45) | 17.9 (10.3)
  M4, Day 31: At 1 hour after morning waketime | 6.80 (2.67) | 14.6 (5.93)
  M9, Day 31: At 1 hour after morning waketime | 1.42 (0.589) | 3.27 (1.50)
  M10, Day 31: At 1 hour after morning waketime | 3.64 (2.17) | 9.04 (5.51)
  Lemborexant, Day 31: At 1.5 hour after morning waketime | 7.40 (4.36) | 17.1 (10.0)
  M4, Day 31: At 1.5 hour after morning waketime | 6.58 (2.76) | 14.1 (5.76)
  M9, Day 31: At 1.5 hour after morning waketime | 1.38 (0.573) | 3.14 (1.46)
  M10, Day 31: At 1.5 hour after morning waketime | 3.67 (2.20) | 8.80 (5.29)

ADVERSE EVENTS:
Time Frame: Run-in Period: From first dose in Run-in Period at Day -14 up to Baseline (Day 1); Treatment Period: From first dose in Treatment Period at Day 1 up to end of follow-up period (up to Day 58)
Groups:
- Run-in Period: Placebo: Participants received one lemborexant-matched PBO tablet, orally, once daily, approximately 5 minutes before intend to sleep for 14 nights from Day -14 up to Baseline (Day 1) during Run-in Period.
- Treatment Period: Placebo: Participants received one lemborexant-matched placebo tablet, orally, once daily, approximately 5 minutes before intend to sleep for 30 nights from Day 1 up to Day 30 in Treatment Period.
- Treatment Period: Lemborexant 5 mg: Participants received one lemborexant 5 mg tablet, orally, once daily, approximately 5 minutes before intend to sleep for 30 nights from Day 1 up to Day 30 in Treatment Period.
- Treatment Period: Lemborexant 10 mg: Participants received one lemborexant 10 mg tablet, orally, once daily, approximately 5 minutes before intend to sleep for 30 nights from Day 1 up to Day 30 in Treatment Period.
Arm/Group | Run-in Period: Placebo | Treatment Period: Placebo | Treatment Period: Lemborexant 5 mg | Treatment Period: Lemborexant 10 mg
All-Cause Mortality (participants affected / at risk) | 0/65 | 0/13 | 0/26 | 0/26
Serious Adverse Events (participants affected / at risk) | 0/65 | 0/13 | 0/26 | 0/26
Other Adverse Events (participants affected / at risk) | 2/65 | 1/13 | 5/26 | 2/26
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Run-in Period: Placebo (N=65) | Treatment Period: Placebo (N=13) | Treatment Period: Lemborexant 5 mg (N=26) | Treatment Period: Lemborexant 10 mg (N=26)
Postural orthostatic tachycardia syndrome (Cardiac disorders) | 0 | 0 | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Oedema peripheral (General disorders) | 0 | 0 | 0 | 1
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Dyslipidaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Arteriosclerosis (Vascular disorders) | 0 | 0 | 0 | 1
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2023-09-14): https://cdn.clinicaltrials.gov/large-docs/89/NCT05594589/Prot_000.pdf
  • Statistical Analysis Plan (2024-07-03): https://cdn.clinicaltrials.gov/large-docs/89/NCT05594589/SAP_001.pdf